CLINICAL TRIAL: NCT02737306
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of PRO 140 for Prophylaxis of Acute Graft-Versus-Host Disease in Patients With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndromes (MDS)
Brief Title: A Study of Acute Graft-Versus-Host Disease (GVHD) in Patients Undergoing Allogeneic Stem-Cell Transplantation
Acronym: GVHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to lack of enrolment..
Sponsor: CytoDyn, Inc. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO 140_CD 03_GVHD
Record Dates: First submitted 2016-03-29; First posted 2016-04-13 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2022-01

CONDITIONS: Graft Vs Host Disease
Keywords: Allogeneic; Stem Cell; Transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — leronlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects were randomized to the blinded part of the study using an IRT system. Unblinded pharmacists at clinical sites were notified of the arm to which the subjects were enrolled in order to prepare the appropriate treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): In this study, 60 subjects will be randomized to receive either PRO 140 or placebo in a 1:1 ratio (i.e. 30 subjects per arm). PRO 140 or placebo will be administered as a 350 mg subcutaneous injection.
  Placebo will be administered -2/-3 days before the stem cell infusion, on the day of stem cell infusion (Day 0) and thereafter on days 7, 14, 21, 28, 42, 56, 70, 84 and 98 as per the study schedule of assessments.
  Each vial of the Placebo contains 5mM Histidine, 15 mM Glycine, 95 mM Sodium Chloride, 0.3% (w/v) Sorbitol, 0.005% (w/v) Polysorbate 20 at a pH of 5.5.
  Each 350 mg dose of placebo consist of 2 SC injections of placebo (5mM Histidine, 15 mM Glycine, 95 mM Sodium Chloride, 0.3% (w/v) Sorbitol, 0.005% (w/v) Polysorbate 20 at a pH of 5.5) of 2 X 1 mL/inj. on opposite sides of abdomen.
  Interventions: Drug: Placebo
- 350 mg Pro140 (Experimental): In this study, 60 subjects will be randomized to receive either PRO 140 or placebo in a 1:1 ratio (i.e.,30 subjects per arm). PRO 140 or placebo will be administered as a 350 mg subcutaneous injection.
  PRO 140 will be administered -2/-3 days before the stem cell infusion, on the day of stem cell infusion (Day 0) and thereafter on days 7, 14, 21, 28, 42, 56, 70, 84 and 98 as per the study schedule of assessments.
  Each vial of the PRO 140 product contains 1.4 mL antibody at 175 mg/ml in a buffer containing 5 mM L-histidine, 15.0 mM glycine, 95 mM sodium chloride, 0.3% (w/v) sorbitol, 0.005% (w/v) polysorbate 20 (Tween 20®), and sterile water for injection, at pH of 5.5.
  Each 350 mg dose of PRO 140 will consist of 2 SC injections of PRO 140 (2 X 1 mL/inj.) on opposite sides of abdomen.
  Interventions: Drug: PRO 140

INTERVENTIONS:
Drug: PRO 140 — PRO 140 is a humanized IgG4,κ monoclonal antibody (mAb) to the chemokine receptor CCR5.
  Other Names: Humanized monoclonal antibody to CCR5
  Arms: 350 mg Pro140
Drug: Placebo — Placebo in parenteral solution.
  Arms: Placebo

SUMMARY:
This is a Phase II, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study of the Safety and Efficacy of PRO 140 for Prophylaxis of Acute Graft-Versus-Host Disease in Patients with Acute Myeloid Leukemia (AML) or Myelodysplastic Syndromes (MDS) Undergoing Allogeneic Stem-Cell Transplantation.

DETAILED DESCRIPTION:
This is a Phase II, randomized, double-blind, placebo-controlled, multi-center study to evaluate the feasibility of the use of PRO 140 as an add-on therapy to standard GVHD prophylaxis treatment for prevention of acute GVHD in adult patients with AML or MDS undergoing allogeneic HCT.

In this study, 60 subjects will be randomized to receive either PRO 140 or placebo in a 1:1 ratio (i.e., 30 subjects per arm). PRO 140 or placebo will be administered as a 350 mg subcutaneous injection on Day -3 or Day -2 prior to stem cell infusion, on the day of stem cell infusion (Day 0), and then weekly for 30 days (at Week 1, Week 2, Week 3 and Week 4) after which it will be administered every two weeks for up to 100±7 days (at Week 6, Week 8, Week 10, Week 12 and Week 14). Subjects will return to clinic for two Follow-up visits at 2 weeks after the last treatment visit, and one year after the first treatment visit.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in the study:

1. Patients diagnosed with AML or MDS per below:

   * Patients with a history of histologically or pathologically confirmed diagnosis of AML and < 5% blasts in the peripheral blood or bone marrow (per bone marrow aspiration and/or biopsy within 6 weeks prior to screening) scheduled to undergo allogeneic stem-cell transplantation
   * Patients with a histologically or pathologically confirmed diagnosis of MDS with < 10% blasts in the bone marrow (per bone marrow aspiration and/or biopsy within 6 weeks prior to screening) scheduled to undergo allogeneic stem-cell transplantation
2. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2
3. Patients must have normal organ function as defined below:

   Myeloablative allogeneic HCT:
   * Males and females, age ≥18 and ≤ 65 years of age
   * Total bilirubin ≤ 2 mg/dL (except in patients with Gilbert's Syndrome)
   * AST/ALT ≤ 3 times institutional upper limit of normal (except in patients with leukemic infiltration of liver)
   * Serum creatinine ≤ 2 mg/dL and creatinine clearance ≥ 60 ml/hr
   * Diffusing capacity of the lung for carbon monoxide (DLCO) > 50% predicted with no symptomatic pulmonary disease
   * Cardiac ejection fraction ≥ 50%. If between 40-49% a cardiology consult is required
   * Clinically normal resting 12-lead ECG at screening visit or, if abnormal, considered not clinically significant by the PI
4. Patients must have a reasonable expectation of ≥ 6 months survival
5. The donor-recipient HLA match criteria required for participation in this protocol are not research subjects in this study and they must meet criteria as National Marrow Donor Program (NMDP) donors. Procedures for selection of donors and stem cell dose will follow FDA requirements for Blood Products (21 CFR 640) and Human Cellular and Tissue Based Products (21 CFR 1271). The standard institutional practices for stem cell transplants also will be followed. The donors are:

   * HLA-Identical Sibling (6/6): Minimal typing necessary is serologic typing for class I (AB) and molecular typing for class II (DRB1)
   * Matched Unrelated Donor (8/8): Molecular identity at HLA A, B, C and DRB1 by high-resolution typing
   * Matched Related and Unrelated Donor (7/8): high-resolution molecular typing at the following loci is required: HLA A, B, C and DRB1
6. Both male and female patients and their partners of childbearing potential must agree to use appropriate birth control methods (birth control pills, barriers, or abstinence) throughout the study duration (excluding women who are not of childbearing potential and men who have been sterilized). Females of childbearing potential must have a negative serum pregnancy test at Screening visit and negative urine pregnancy test prior to receiving the first dose of study drug.
7. Patients must understand and voluntarily sign an informed consent form

Exclusion Criteria

Subjects meeting any of the following criteria will be excluded from the study:

1. Patients not expected to be available for follow-up for at least 114 days after transplant
2. Patients who have received prior allogeneic stem cell-transplantation
3. Patients who receive post-transplant high dose cyclophosphamide
4. Patients with active central nervous system (CNS) involvement by malignant cells
5. Patients receiving other investigational drugs for GVHD. Co-enrollment in other clinical trials that do not include experimental GVHD therapies is allowed.
6. Prior use of any experimental or approved CCR5 modulator including maraviroc and PRO 140
7. Patients with uncontrolled bacterial, viral or fungal infections including diagnosis of acute viral hepatitis (defined as any active infection with hepatitis A or a new diagnosis of hepatitis B or C within 24 weeks of dosing)
8. Currently active second malignancy other than non-melanoma skin cancers
9. Presence of fluid collection (ascites, pleural or pericardial effusion) that interferes with methotrexate clearance or makes methotrexate use contraindicated
10. Patients who are HIV positive
11. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study
12. Subjects on chronic steroid therapy > 5 mg/day within 2 weeks of screening except for inhaled, nasal, or topical steroids
13. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-05-14 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Loyola University Medical Center Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Transplant Institute Methodist Hospital, San Antonio, Texas
  - West Virginia University Medicine, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PRO 140: In this study, 60 subjects will be randomized to receive either PRO 140 or placebo in a 1:1 ratio (i.e. 30 subjects per arm). PRO 140 or placebo will be administered as a 350 mg subcutaneous injection on Day -3 or Day -2 prior to stem cell infusion, on the day of stem cell infusion (Day 0), and then weekly for 30 days (at Week 1, Week 2, Week 3 and Week 4) after which it will be administered every two weeks for up to 100±7 days (at Week 6, Week 8, Week 10, Week 12 and Week 14). Subjects will return to clinic for two Follow-up visits at 2 weeks after the last treatment visit, and one year after the first treatment visit.
  PRO 140: Two 1 mL injections, 175mg/ml each, of PRO 140 to opposite sides of the abdomen.
- Placebo: In this study, 60 subjects will be randomized to receive either PRO 140 or placebo in a 1:1 ratio (i.e. 30 subjects per arm). PRO 140 or placebo will be administered as a 350 mg subcutaneous injection on Day -3 or Day -2 prior to stem cell infusion, on the day of stem cell infusion (Day 0), and then weekly for 30 days (at Week 1, Week 2, Week 3 and Week 4) after which it will be administered every two weeks for up to 100±7 days (at Week 6, Week 8, Week 10, Week 12 and Week 14). Subjects will return to clinic for two Follow-up visits at 2 weeks after the last treatment visit, and one year after the first treatment visit.
  Placebo: Two 1 mL injections, 175mg/ml each (placebo contains 5mM Histidine, 15 mM Glycine, 95 mM Sodium Chloride, 0.3% (w/v) Sorbitol, 0.005% (w/v) Polysorbate 20 at a pH of 5.5) to opposite sides of the abdomen.
Period: Overall Study
Arm/Group | PRO 140 | Placebo
Started | 6 | 5
Completed | 2 | 5
Not Completed | 4 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Enrolment and treatment halted by sponsor. | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population is defined as the set of subjects who are randomized to PRO 140 or placebo. The ITT population will be the primary analysis population for the analysis of primary and secondary endpoints
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO 140 | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 43 [25 to 61] | 54 [39 to 63] | 48 [25 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11
HIV rapid antigen test [Count of Participants; unit: Participants]
  HIV rapid antigen test negative | 6 | 5 | 11
  HIV rapid antigen test positive | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute GVHD by Day 100
Description: Incidence of Grade II, Grade III or Grade IV acute GVHD by Day-100
Time Frame: 100 days from first treatment (100 Days post treatment)
Population: Study was terminated before outcome data could be obtained.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence of Severe and Life-threatening (Grade III and Grade IV) Acute GVHD by Day-100
Description: The number and percentages of subjects with severe and life-threatening (Grade III and Grade IV) acute GVHD by Day-100 will be presented. Chi-square/ Fisher's exact test will be used to compare the incidence between the treatment groups.
Time Frame: 100 Days post-treatment
Population: Study was terminated before secondary efficacy endpoint data could be obtained.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Organ-specific Acute GVHD by Day-100
Description: The number and percentages of subjects with organ-specific acute GVHD by Day-100 will be presented by organ category. Chi-square/ Fisher's exact test will be used to compare the incidence between the treatment groups.
Time Frame: 100 Days post-treatment
Population: Study was terminated before secondary efficacy endpoint data could be obtained.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Donor Engraftment Evaluated by T-cell and Myeloid Chimerism in Peripheral Blood
Description: The number and percentages of subjects with donor engraftment failure evaluated by T-cell and myeloid chimerism in peripheral blood will be presented by different treatment groups. Chi-square/ Fisher's exact test will be used to compare the incidence of donor engraftment failure.
Time Frame: 365 days post-initial treatment (T1 Visit) (+/- 14 days)
Population: Study was terminated before secondary efficacy endpoint could be obtained.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Neutrophil and Platelet Count Recovery
Description: The number and percentages of subjects with neutrophil and platelet count recovery will be presented. Chi-square/ Fisher's exact test will be used to compare the incidence of neutrophil recovery and of platelet recovery between treatment groups.
Time Frame: 100 Days post treatment
Population: Study was terminated before secondary endpoint data could be obtained.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Changes in ECOG Performance Score
Description: The raw and change from baseline in ECOG performance score will be summarized for each assessment scheduled visit (i.e., Screening visit, Treatment Visits 1, 4, 7, 9, 11, Follow-up Visit 1and Unscheduled Visit(s)). Descriptive statistics (n, mean, standard deviation, median, minimum and maximum) will be presented by treatment group. If the Normality assumption is met, t-test will be used to compare the mean of ECOG performance score between the treatment groups and if the Normality assumption is not met, a non-parametric method will be used.
Time Frame: 100 Days post treatment visit 1
Population: Trial was terminated before secondary endpoint data could be obtained.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: GVHD-free Survival (GFS)
Description: GFS will be defined as the elapsed time between the date of transplant until GVHD related death. GVHD-free survival will be compared between the treatment groups using Log-rank test and Kaplan-Meier methods will be used to depict the survival curves.
Time Frame: 100 Days post treatment visit T1
Population: Study was terminated before secondary efficacy endpoint data could be obtained.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Tolerability of Repeated Subcutaneous Administration of PRO 140 as Assessed by Study Participants (Using Visual Analogue Scale) and by Investigator-evaluation of Injection Site Reactions
Description: All data from tolerability assessments of repeated subcutaneous administration of PRO 140 as assessed by study participants and by investigator-evaluation of injection site reactions will be summarized using n, mean, Standard Deviation (SD), minimum and maximum values.
Time Frame: 365 days post-treatment (+/- 14 days)
Population: Study was terminated before secondary efficacy endpoint data could be obtained.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Frequency of Treatment Emergent Adverse Events and Serious Adverse Events
Description: Frequency of treatment emergent adverse events and treatment emergent serious adverse events.
Time Frame: 100 Days post treatment
Population: Study was terminated before secondary efficacy endpoint data could be obtained.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: AML or MDS Relapse Rate by Day-100
Description: AML or MDS relapse rate by Day-100 will be summarized and present by treatment groups.
Time Frame: 100 Days post treatment
Population: Study was terminated before secondary efficacy endpoint data could be obtained.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Changes and Shifts in Laboratory Measurements Over Time
Description: Safety Assessment- The laboratory measurements will include Routine CBC, Biochemistry and Urinalysis.
  * Routine CBC includes hemoglobin, hematocrit (HCT), red blood cell (RBC) count, white blood cell (WBC) count, WBC differential count (%), absolute neutrophils count (ANC) and platelets count.
  * Biochemistry profile includes assessment of Hepatic function indicators: total and direct bilirubin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), total protein, Lactate dehydrogenase (LDH); Renal function indicators: Blood Urea Nitrogen (BUN), creatinine; Electrolytes: sodium, potassium, chloride, calcium and bicarbonate; Other: glucose (random), cholesterol (total)
  * Urinalysis for color, appearance, specific gravity, pH, protein, glucose, occult blood, ketones, RBC, WBC, epithelial cells, bacteria, casts, crystals
Time Frame: 365 days post-treatment (+/- 14 days)
Population: Trial was terminated before outcome measure data could be obtained.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Changes in Electrocardiogram (ECG) Parameters Over Time
Description: Safety Assessment-The following ECG parameters will be evaluated: ventricular rate (beats per minute), PR interval (msec), QRS interval (msec), QT interval (msec), and QTc interval (msec).
Time Frame: 365 days post-treatment (+/- 14 days)
Population: Trial was terminated before secondary outcome measure data was obtained.
Arm/Group | PRO 140 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: Adverse events were systematically assessed through documented symptom-directed physical examinations, vital sign evaluation and injection site reaction evaluations performed at treatment and follow-up visits. All information is collected on case report forms.
Arm/Group | PRO 140 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 6/6 | 1/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRO 140 (N=6) | Placebo (N=5)
Acute graft versus host disease (Immune system disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pyrexia (General disorders) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRO 140 (N=6) | Placebo (N=5)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
Dry eye (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 | 0
Apoptotic colonopathy (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 2
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Oral blood blister (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2
Asthenia (General disorders) | 1 | 0
Catheter site bruise (General disorders) | 1 | 0
Catheter site erythema (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 3
Infusion site pruritus (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 2 | 3
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 1
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Acute graft versus host disease (Immune system disorders) | 1 | 0
Graft versus host disease (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Serum sickness (Immune system disorders) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Viraemia (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Vulvovaginal injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 2 | 3
International normalised ratio increased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 4 | 3
Platelet count decreased (Investigations) | 2 | 5
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 4 | 2
Lethargy (Nervous system disorders) | 1 | 1
Lhermitte's sign (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Taste disorder (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vulval oedema (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngeal lesion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Sinus operation (Surgical and medical procedures) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 2 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
Superficial vein thrombosis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was stopped prior to completion due to lack of enrolment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT02737306/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT02737306/SAP_001.pdf